CLINICAL TRIAL: NCT01562119
Title: Long Term Evaluation of Human Acellular Dermal Matrix Allograft For Coverage of the Wound After Extensive Deep Burn
Acronym: ADM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Xiaolin Wang，Principal Investigator, Ms., Tang-Du Hospital
Other Study IDs: TDLL-2012109
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Burn; Traumatic Implants
Keywords: Burns; Wound repair; Skin substitutes
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The skin with ADM inplant and the nomal skin as control group
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The present study was to retrospectively evaluate the long-term outcomes of the cograft acellular dermal matrix (ADM) with autologous thin split-thickness skin for coverage of functional regional wounds in burned patients.

DETAILED DESCRIPTION:
The potential of acellular dermal matrix (ADM) had been proved to improve cosmetic and functional outcomes, nevertheless, there had been few reports about the long term results of the morphological, histological and functional changes after placement. The present study was to retrospectively evaluate the long-term outcomes of the cograft acellular dermal matrix (ADM) with autologous thin split-thickness skin for coverage of functional regional wounds in burned patients.

ELIGIBILITY:
Inclusion Criteria:

* the patient's skin with ADM implant

Exclusion Criteria:

Ages: 3 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Thirty burn patients, treated by composite graft of ADM with autologous split-thickness skin from January 2007 to December 2009, were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Function of the region covered by human acellular dermal matrix allograft | March, 2012 to May, 2013

SECONDARY OUTCOMES:
Physical characteristics of the transplanted human acellular dermal matrix allograft | March, 2012 to May, 2013

CONTACTS AND LOCATIONS:
Overall Officials: Xueyong Li, Doctor, Study Director — Department of Burn and Plastic Sugery
Locations (1):
- Department of Burn and Plastic Sugery, Tangdu Hospital, Xi'an, Shaanxi, China